CLINICAL TRIAL: NCT02611128
Title: Urinary DENND1A.V2 as a Predictor of Pubertal Hyperandrogenemia
Acronym: DENND1A
Status: Suspended | Type: Observational
Why Stopped: temporarily closed to enrollment due to COVID
Sponsor: University of Virginia (Other)
Collaborators: Penn State University (Other); Virginia Commonwealth University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chris McCartney, Associate Professor of Medicine, University of Virginia
Other Study IDs: 17633; P50HD028934 (NIH)
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Polycystic Ovary Syndrome; Hyperandrogenism; Puberty
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Phenotype

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Optional sample banking for later genetic analysis: At the time of study, the investigators will request consent/assent to bank saliva samples for later genetic analysis (e.g., if additional highly-promising gene candidates for adolescent hyperandrogenemia/PCOS are identified). If subjects and parents do not provide assent/consent that would allow specimens to be banked for later genetic analysis, the samples and the means of linking specimens to data will be destroyed (once analysis for all participants is completed).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peripubertal girls: Peripubertal girls with varying androgen concentrations will have careful phenotype/genotype assessment, primarily to assess the relationship between urinary exosomal DENND1A.V2 and serum free testosterone concentrations.
  Interventions: Other: Phenotype/genotype assessment

INTERVENTIONS:
Other: Phenotype/genotype assessment — The investigators will perform careful phenotyping in addition to hormonal assessments and assessments of DENND1A

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common disorder marked by hyperandrogenism, oligo-/anovulation, and subfertility. The precise causes of PCOS are unclear, but the pathophysiology involves complex genetic and environmental influences. Importantly, not all girls with obesity have HA, and free testosterone (T) concentrations are highly variable in this group. Luteinizing hormone (LH) and insulin concentrations are significant but only partial predictors of free T in girls with obesity; significant unexplained variability in free T suggests that additional factors contribute to HA in this population. Abnormalities of ovarian and adrenal steroidogenesis are likely contributors in this regard, but such abnormalities are difficult to quantify. Recent Genome Wide Association Studies have identified DENND1A as a PCOS susceptibility gene candidate. Preliminary in vitro data strongly implicate a DENND1A splice variant called DENND1A Variant 2 (DENND1A.V2) as a contributor to excessive theca cell androgen production in PCOS. The investigators' primary goal with the proposed pilot study is to determine the relationship between urinary exosomal DENND1A.V2 mRNA and free T concentrations in peripubertal girls. The investigators hypothesize that urinary exosomal DENND1A.V2 mRNA quantity is a significant and independent predictor of peripubertal hyperandrogenemia. In this study, the investigators will carefully phenotype peripubertal girls with and without hyperandrogenemia (primarily in the form of hormonal, maturational, and anthropometric measurements) in addition to measuring urinary exosomal DENND1A.V2 mRNA. As a primary analysis, the investigators will examine the relationship between morning free testosterone and urinary exosomal DENND1A.V2, controlling for previously-described partial predictors of free testosterone (LH, insulin) in addition to potential confounders (BMI z-score, bone age). These studies will provide important information regarding the etiology of HA in peripubertal girls. Ultimately, these data may lead to a non-invasive test of ovarian/adrenal steroidogenic activity and support the development of a diagnostic test for PCOS in high-risk peripubertal girls (e.g., those with obesity).

DETAILED DESCRIPTION:
To date, the mechanisms underlying excess androgen production from steroid producing tissues have been unclear, but recent Genome Wide Association Studies (GWAS) have provided additional data in this regard. Initial GWAS data in a Han Chinese population identified some 12 loci as potential PCOS susceptibility gene candidates. One of these loci, the DENND1A locus at 9q22.32, has been replicated in GWAS studies in both Asian and European populations. Strauss and colleagues recently demonstrated DENND1A expression in testes, ovarian theca cells, and H295 adrenal carcinoma cells - all androgen producing tissues/cells. DENND1A is therefore an exceedingly strong PCOS susceptibility gene candidate. However, it remains unclear how DENND1A may contribute to the PCOS phenotype.

Importantly, there are two transcriptional forms of the DENND1A gene - a consequence of alternate splicing. The larger transcript (DENND1A Variant 1, or DENND1A.V1) encodes a 1009 amino acid protein, while the smaller transcript DENND1A.V2 encodes a truncated 559 amino acid. The product of DENND1A.V2 contains the DENN domain and a clathrin-binding domain, but differs from the product of DENND1A.V1 in two ways: (1) it does not contain the proline-rich C-terminal domain present in Variant 1, and (2) DENND1A.V2 results from differential splicing and contains a unique 33 amino acid C-terminal sequence. Of significant interest, published studies by Drs. McAllister and Strauss (McAllister JM, et al. Proc Natl Acad Sci USA. 2014;111:E1519-27) strongly implicate the DENND1A.V2 splice variant as a contributor to excessive theca cell androgen production in PCOS:

* Expression of DENND1A.V2 protein in cultured theca cells isolated from women with PCOS was over 3-fold elevated compared to normal ovarian theca cells. Similarly, DENND1A.V2 mRNA abundance was elevated in PCOS theca and correlated with increased theca cell androgen (dehydroepiandrosterone [DHEA]) production.
* Forced expression of DENND1A.V2 in normal theca cells increased expression of CYP17A1 and CYP11A1 (genes for key steroidogenic enzymes) along with androgen/androgen precursor (e.g., 17OHP4, DHEA, testosterone) and progesterone production.
* Knockdown of DENND1A.V2 in cultured PCOS theca cells reduced CYP17A1 and CYP11A1 expression in addition to 17OHP4 and DHEA production.
* Treatment of cultured PCOS theca cells with anti-DENND1A.V2 IgG antibodies reduced expression of CYP17A1 and CYP11A1 mRNA expression as well as DHEA and 17OHP4 synthesis.

These data provide strong support to the contention that the DENND1A.V2 splice variant is a major factor underlying the phenotype of cultured PCOS theca cells and, thus, the etiology of ovarian hyperandrogenemia in PCOS. By extension, the DENND1A.V2 splice variant may be a significant contributor to peripubertal hyperandrogenemia, and it may explain much of the variable hyperandrogenemia observed in obese peripubertal girls. The investigators propose that, in some peripubertal girls, increased expression of DENND1A.V2 in ovarian and/or adrenal cells promotes excess androgen secretion with the advent of puberty (when ovarian stimulation by LH increases) and/or in the presence of obesity (e.g., enhanced insulin secretion, augmenting LH-stimulated ovarian androgen synthesis and/or ACTH-stimulated adrenal androgen synthesis).

Of great interest, preliminary data from 5 normal women and 6 women with PCOS suggested that urinary exosomal DENND1A.V2 mRNA was approximately 3-fold elevated in women with PCOS compared to normally-cycling controls (McAllister JM, et al. Proc Natl Acad Sci USA. 2014;111:E1519-27). Exosomes are small vesicles (40-100 nm) that contain nucleic acids shed by cells into blood and urine, and they are known to be a stable source of RNA. Thus, urinary exosomal DENND1A.V2 quantity may serve as a marker of DENND1A.V2 activity in the ovary/adrenal.

In these proposed studies, the investigators (including collaborators Drs. McAllister and Strauss) will obtain urine for exosomal DENND1A.V2 mRNA quantitation in addition to blood samples to measure androgen levels, LH and insulin (the latter two previously-demonstrated to predict free testosterone). The investigators will test the hypothesis that the quantity of urinary exosomal DENND1A.V2 mRNA is a strong and independent predictor of androgen levels in peripubertal girls.

To the investigators' knowledge, no data exist that tie a PCOS susceptibility gene candidate to pubertal hyperandrogenemia. The investigators propose to evaluate a novel biomarker (urinary exosomal DENND1A.V2 mRNA) as a predictor of free testosterone in pubertal girls. Evaluation of this biomarker in adolescents is highly innovative.

The present proposal will build on Aim 3 of Project 1 (NIH P50 HD28934), in which the investigators carefully assess the determinants of hyperandrogenemia in girls with peripubertal obesity. Specifically, Aim 3 is an intensive protocol involving (a) overnight frequent blood sampling for LH and insulin along with (b) ovarian and adrenal stimulation protocols over the subsequent 2 days. Some of the subjects participating in this proposed pilot study will also participate in Aim 3. Correlation between urinary exosomal DENND1A.V2 mRNA and ovarian/adrenal stimulation protocols will allow a preliminary assessment of urinary exosomal DENND1A.V2 mRNA as a non-invasive measure of ovarian/adrenal steroidogenesis - a potentially important clinical tool.

Peripubertal girls with hyperandrogenemia are believed to be at high risk for developing adolescent/adult PCOS, but since the manifestations of PCOS can overlap with the findings of normal puberty, the diagnosis of PCOS may be unreliable until later adolescence. If urinary exosomal DENND1A.V2 mRNA is a significant predictor of hyperandrogenemia in this cohort, future studies will determine the utility of urinary exosomal DENND1A.V2 as a diagnostic test to predict the development of PCOS across puberty. This is an innovative and exceedingly exciting prospect that may have significant potential implications for at-risk girls.

ELIGIBILITY:
List of Inclusion Criteria

• Peripubertal girls, Tanner breast stages 1-5

List of Exclusion Criteria

* Age < 8 or > 17 y
* Men and boys are excluded
* Inability to obtain proper consent/assent
* Atypical obesity
* Underweight: Underweight is defined as a BMI-for-age percentile < 5
* Positive pregnancy test or lactation
* Assessment during the luteal phase as suggested by a serum progesterone ≥ 1.5 ng/ml
* Virilization or a total testosterone > 150 ng/dl
* Excessively elevated DHEA-S: This will be defined as a DHEA-S > 1.5 times the age-appropriate upper limit of normal
* Congenital adrenal hyperplasia (CAH)
* Cortisol deficiency/excess
* Inadequately-treated or unstable thyroid dysfunction
* Significant hyperprolactinemia: Since mild elevations may be seen in girls with hyperandrogenemia or PCOS, elevations up to 30 (i.e., 1.5 times the upper limit of normal) will be accepted in such girls
* Significant chronic medical history: This includes a significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; asthma requiring intermittent systemic corticosteroids; etc.); history of renal insufficiency or durable electrolyte abnormalities; or a history of substantial liver disease. A history of liver test abnormalities will be allowed in two circumstances: (1) mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome; (2) mild transaminase (ALT, AST) elevations may be seen in obese girls, so stable elevations < 1.5 times the upper limit of normal will be accepted in this group.
* Uncontrolled type 2 diabetes mellitus: This will be reflected by a hemoglobin A1c > 7.0%. Subjects with impaired glucose tolerance or a diagnosis of type 2 diabetes that is well-controlled with lifestyle management alone will be allowed to participate.
* Type 1 diabetes mellitus: Since subjects with type 1 diabetes invariably require exogenous insulin, they will not be allowed to participate.

Ages: 8 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Peripubertal girls, Tanner breast stages 1-5
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2015-05-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Urinary exosomal DENND1A.V2 | Day 1 of study (the study involves one outpatient visit)
  Urinary exosomal DENND1A.V2
Serum free testosterone | Day 1 of study (the study involves one outpatient visit)
  Calculated free testosterone

SECONDARY OUTCOMES:
Bone age | Day 1 of study (the study involves one outpatient visit)
  A measure of maturational stage
BMI z-score | Day 1 of study (the study involves one outpatient visit)
  Body mass index normalized for age and gender
Morning luteinizing hormone | Day 1 of study (the study involves one outpatient visit)
  Serum luteinizing hormone (LH) measured at same time as free testosterone and fasting insulin
Fasting insulin | Day 1 of study (the study involves one outpatient visit)
  Serum insulin measured at same time as free testosterone and morning LH

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- Center for Research in Reproduction, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not have current plans to share IPD